CLINICAL TRIAL: NCT04432584
Title: A Phase III, Randomized, Open-label, Active-controlled, Multicenter Study Evaluating the Safety, Pharmacokinetics, Pharmacodynamic and Efficacy of Crovalimab Versus Eculizumab in Patients With Paroxysmal Nocturnal Hemoglobinuria (PNH) Currently Treated With Complement Inhibitors
Brief Title: A Study Evaluating the Safety, Pharmacokinetics, and Efficacy of Crovalimab Versus Eculizumab in Participants With Paroxysmal Nocturnal Hemoglobinuria (PNH) Currently Treated With Complement Inhibitors
Acronym: COMMODORE 1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO42161; 2020-000597-26 (EudraCT Number); 2023-506526-37-00 (EU CTIS Number)
Record Dates: First submitted 2020-06-03; First posted 2020-06-16 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Crovalimab) (Experimental): Participants will receive a loading series of crovalimab comprised of an intravenous (IV) dose on Day 1, followed by weekly crovalimab subcutaneous (SC) doses for 4 weeks on Week 1 Day 2, then on Weeks 2, 3, and 4. Maintenance SC dosing will begin at Week 5 and will continue every 4 weeks (Q4W) thereafter for a total of 24 weeks of study treatment. After 24 weeks of crovalimab treatment, participants who derive benefit from the drug may continue to receive crovalimab.
  Interventions: Drug: Crovalimab
- Arm B (Eculizumab) (Active Comparator): Participants will receive an approved maintenance dose of eculizumab starting on Day 1 and every 2 weeks (Q2W) thereafter for a total of 24 weeks of study treatment. After 24 weeks of study eculizumab treatment, participants will have the option to switch to crovalimab or to discontinue from the study after completion of 10 weeks of safety follow-up.
  Interventions: Drug: Eculizumab
- Arm C (Crovalimab) (Exploratory) (Experimental): Participants with a body weight ≥ 5 to <12 kilograms (kg) will receive a loading series of crovalimab doses comprised of an IV dose on Day 1 of Week 1, followed by crovalimab SC dose on Day 2 Week 1. Maintenance doses will begin at Week 3 and will be administered Q2W, thereafter. Participants with a body weight ≥ 12 to < 20 kg and ≥ 20 kg will receive a loading series of crovalimab doses comprised of an IV dose on Day 1 of Week 1, followed by weekly crovalimab SC doses for 4 weeks at Week 1 (Day 2) and then at Weeks 2, 3, and 4. Maintenance doses will begin at Week 5 and will be administered Q2W thereafter, for participants with a body weight ≥ 12 to < 20 kg and Q4W thereafter, for participants with a body weight > 20 kg. After 24 weeks of crovalimab treatment, participants who derive benefit from the drug may continue to receive crovalimab.
  Interventions: Drug: Crovalimab

INTERVENTIONS:
Drug: Crovalimab — Dosing depends on body weight. Participants will be dosed as follows:
  * 5 kg to < 12 kg: 100 mg IV on Week 1 Day 1 (W1D1); 85 mg SC on Week 1 Day 2 (W1D2) and Q2W from Week 3 until end of study
  * 12 kg to < 20 kg: 200 mg IV on W1D1; 85 mg SC on W1D2, Weeks 2, 3 and 4; 170 mg SC, Q2W from Week 5 until end of study
  * 20 kg to < 30 kg: 300 mg IV on W1D1; 85 mg SC on W1D2, Weeks 2, 3 and 4; 340 mg SC, Q4W from Week 5 until end of study
  * 30 kg to < 40 kg: 400 mg IV on W1D1; 170 mg SC on W1D2, Weeks 2, 3 and 4; 510 mg SC, Q4W from Week 5 until end of study
  * 40 kg to < 100 kg: 1000 mg IV on W1D1; 340 mg SC W1D2, Weeks 2, 3 and 4; 680 mg SC, Q4W from Week 5 until end of study
  * 100 kg: 1500 mg IV on W1D1; 340 mg SC W1D2, Weeks 2, 3 and 4; 1020 mg SC, Q4W from Week 5 until end of study.
  Arms: Arm A (Crovalimab); Arm C (Crovalimab) (Exploratory)
Drug: Eculizumab — Eculizumab will be administered at a dose of 900 mg Q2W, as per the dosing schedule described above.
  Arms: Arm B (Eculizumab)

SUMMARY:
A study designed to evaluate the safety of crovalimab with eculizumab in participants with PNH currently treated with complement inhibitors. This study will enroll approximately 190 participants.

ELIGIBILITY:
Inclusion Criteria:

* Body weight ≥ 40 kg at screening (pediatric participants with body weight < 40 kg)
* Treated with eculizumab or ravulizumab for PNH for at least 3 months prior to Day 1
* Lactate Dehydrogenase Levels ≤ 2x the upper limit of normal (ULN) at screening
* Willingness and ability to comply with all study visits and procedures
* Documented diagnosis of PNH, confirmed by high sensitivity flow cytometry
* Vaccination against Neisseria meningitidis serotypes A, C, W, and Y < 3 years prior to initiation of study treatment; or, if not previously done, vaccination administered no later than one week after the first drug administration
* Women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception during the treatment period and for 10.5 months after the final dose of crovalimab or for 3 months after the final dose of eculizumab (or longer if required by the local product label)

Exclusion Criteria:

* History of allogeneic bone marrow transplantation
* History of myelodysplastic syndrome with Revised International Prognostic Scoring System (IPSS-R) prognostic risk categories of intermediate, high and very high
* Pregnant or breastfeeding, or intending to become pregnant during the study, within 10.5 months after the final dose of crovalimab, or 3 months after the final dose of eculizumab (or longer if required by the local product label)
* Participation in another interventional treatment study with an investigational agent or use of any experimental therapy within 28 days of screening or within 5 half-lives of that investigational product, whichever was greater: participants enrolled in an eculizumab or ravulizumab interventional study are eligible provided they fulfill eligibility (e.g., are willing and able to comply with the study assessments) and stop their participation in current trial before randomisation/enrolment
* Positive for Active Hepatitis B and C infection (HBV/HCV)
* Concurrent disease, treatment, procedure, or surgery or abnormality in clinical laboratory tests that could interfere with the conduct of the study, may pose any additional risk for the participant, or would, in the opinion of the investigator, preclude the participant's safe participation in and completion of the study
* History of or ongoing cryoglobulinemia at screening

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2020-09-30 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) and by Severity | Up to approximately 6 years
  Severity determined according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events, Version 5 (CTCAE v5).
Percentage of Participants With Injection-site Reactions, Infusion-related Reactions, Hypersensitivity and Infections (including Meningococcal Meningitis) | Up to approximately 6 years
Percentage of Participants With Adverse Events (AEs) Leading to Study Drug Discontinuation | Up to approximately 6 years
Percentage of Participants With Clinical Manifestations of Drug-target-drug Complex (DTDC) Formation Amongst Those Participants Who Switched to Crovalimab Treatment From Eculizumab Treatment or Ravulizumab Treatment | Up to approximately 6 years

SECONDARY OUTCOMES:
Serum Concentrations of Crovalimab or Eculizumab Over Time | Up to approximately 6 years
Serum Concentrations of Ravulizumab at the Time of Crovalimab Initiation | Baseline
Percentage of Participants With Anti-crovalimab Antibodies | Up to approximately 6 years
Change in Pharmacodynamic (PD) Biomarker Complement Activity (CH50) Over Time | Up to approximately 6 years
Change Over Time in Free C5 Concentration in Crovalimab-treated Participants | Up to approximately 6 years
Observed Value in Reticulocyte Count (count/milliliters [mL]) | Up to approximately 6 years
Observed Value in Free Hemoglobin and Haptoglobin (milligrams per deciliter [mg/dL]) | Up to approximately 6 years
Absolute Change From Baseline in Reticulocyte Count (count/mL) | Baseline up to Week 25
Absolute Change From Baseline in Free Hemoglobin and Haptoglobin (mg/dL) | Baseline up to Week 25

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (81):
- United States (2):
  - Carolinas Healthcare System, Charlotte, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
- Belgium (3):
  - Cliniques Universitaires Saint-Luc, Brussels
  - AZ Delta Campus Westlaan, Roeselare
  - CHU UCL Namur / site Godinne, Yvoir
- Brazil (9):
  - Chronos Pesquisa Clinica, Taguatinga, Federal District
  - Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital de Clínicas de Porto Alegre X, Porto Alegre, Rio Grande do Sul
  - Instituto Joinvilense de Hematologia E Oncologia, Joinville, Santa Catarina
  - Hospital das Clínicas FMRP-USP, Ribeirão Preto, São Paulo
  - *X*CEPHO - Centro de Estudos e Pesquisas em Hematologia e Oncologia, Santo André, São Paulo
  - Hospital Sírio-Libanês, São Paulo, São Paulo
  - Hospital Paulistano, São Paulo, São Paulo
  - Beneficencia Portuguesa de Sao Paulo, São Paulo
- Ustav hematologie a krevni transfuze, Prague, Czechia
- North Estonia Medical Centre Foundation, Tallinn, Estonia
- Hopital Claude Huriez - CHU Lille, Lille, France
- Germany (2):
  - Universitaetsklinikum Aachen AOeR, Aachen
  - ELBLANDKLINIKUM Riesa, Riesa
- Greece (2):
  - General Hospital of Athens LAIKO, Athens
  - Attikon University General Hospital, Athens
- Prince of Wales Hospital, Hong Kong, Hong Kong
- Semmelweis Egyetem, Budapest, Hungary
- St James's Hospital, Dublin, Ireland
- Italy (5):
  - Azienda Unita Sanitaria Locale- Ravenna, Ravenna, Emilia-Romagna
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Lazio
  - Fondazione IRCCS CA? Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Turin, Piedmont
  - Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
- Japan (15):
  - Fujita Health University Hospital, Aichi
  - Kobe University Hospital, Hyōgo
  - Tokushukai Takasago Seibu Hospital, Hyōgo
  - Ishikawa Prefectural Central Hospital, Ishikawa
  - Tokai University Hospital, Kanagawa
  - Mie University Hospital, Mie
  - Japanese Red Cross Society Suwa Hospital, Nagano
  - Nagasaki University Hospital, Nagasaki
  - Sasebo City General Hospital, Nagasaki
  - National Hospital Organization Okayama Medical Center, Okayama
  - The University of Osaka Hospital, Osaka
  - Iwate Prefectural Isawa Hospital, Ōshū
  - NTT Medical Center Tokyo, Tokyo
  - Tokyo Medical University Hospital, Tokyo
  - Toyama Prefectual Central Hospital, Toyama
- Amsterdam UMC, Locatie AMC, Amsterdam, Netherlands
- Poland (5):
  - Szpital Uniwersytecki nr2 im. dr J. Biziela, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Gda?sk
  - Samodzielny Publiczny Szpital Kliniczny nr 1, Lublin
  - Pratia Poznan, Skórzewo
  - MTZ Clinical Research Powered by Pratia, Warsaw
- Portugal (2):
  - Centro Hospitalar do Baixo Vouga E.P.E. - Hospital de Aveiro, Aveiro
  - Centro Hospitalar do Porto - Hospital de Santo António, Porto
- King Faisal Specialist Hospital & Research Center, Riyadh, Saudi Arabia
- National University Hospital, Singapore, Singapore
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Ulsan University Hospital, Ulsan
- Spain (12):
  - ICO Badalona - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Complejo Hospitalario Universitario de Santiago., Santiago de Compostela, LA Coruna
  - Hospital U. Central de Asturias, Asturias, Principality of Asturias
  - Hospital de Basurto, Bilbao, Vizcaya
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Clinico San Carlos, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario de Toledo, Toledo
  - Hospital Universitario Miguel Servet, Zaragoza
- Akademiska Sjukhuset, Uppsala, Sweden
- Taiwan (3):
  - Changhua Christian Hospital, Chang-hua
  - Hualien Tzu Chi Hospital, Hualien City
  - National Taiwan Universtiy Hospital, Taipei
- Turkey (Türkiye) (6):
  - Hacettepe University Medical Faculty; Neurology, Ankara
  - Gaziantep University Medical Faculty Sahinbey Educational Research Hospital; Hematology, Gaziantep
  - Istanbul University Istanbul Medical Faculty; Neurology, Istanbul
  - Marmara University Pendik Training and Research Hospital, Hematology Department, Istanbul
  - Ege University Medical Faculty; Hematology, Izmir
  - Ondokuz Mayis Univ. Med. Fac., Samsun
- King'S College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Kulasekararaj AG, Nishimura JI, Roth A, Beveridge L, Buatois S, Buri M, Compagno N, Luder Y, Sreckovic S, Scheinberg P. Managing transient immune complex reactions in patients with paroxysmal nocturnal hemoglobinuria: clinical observations from the COMMODORE 1 and 2 studies. Ther Adv Hematol. 2025 Sep 17;16:20406207251359246. doi: 10.1177/20406207251359246. eCollection 2025. PMID 40978458
- [Derived] Roth A, Fu R, He G, Alzahrani H, Chou SC, Hicheri Y, Kazmierczak M, Recova VL, Uchiyama M, Vladareanu AM, Beveridge L, Buatois S, Buri M, Compagno N, Shi D, Balachandran N, Sreckovic S, Scheinberg P. Safety of Crovalimab Versus Eculizumab in Patients With Paroxysmal Nocturnal Haemoglobinuria (PNH): Pooled Results From the Phase 3 COMMODORE Studies. Eur J Haematol. 2025 Feb;114(2):373-382. doi: 10.1111/ejh.14339. Epub 2024 Nov 13. PMID 39535306